CLINICAL TRIAL: NCT04694027
Title: Omega-3 Fatty Acids Plus Vitamin E Cosupplementation Versus Vitamin E in Fibrocystic Breast Patient
Acronym: FCC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rehab Sabry, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Omega 3 & vit E for mastalgia
Record Dates: First submitted 2020-12-31; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Mastalgia
MeSH Terms: conditions — Mastodynia | interventions — Fatty Acids, Omega-3; Tocopherols

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group a (Active Comparator): will receive omega 3 plus vitamin E
  Interventions: Drug: Omega 3 fatty acid; Drug: VitaE
- Group b (Active Comparator): will receive vitamin E
  Interventions: Drug: VitaE
- Group c (No Intervention): no intervention just reassurance and analgesics on need

INTERVENTIONS:
Drug: Omega 3 fatty acid — omega 3 1000 mg
  Arms: group a
Drug: VitaE — vitamin e 400 mg
  Arms: Group b; group a

SUMMARY:
to identify the effect of omega-3 plus vitamin E cosupplementation on mastalgia in patients with FCC and to compare its effect with that of vitamin E only.

DETAILED DESCRIPTION:
120 patients will be enrolled in the study and divided into three groups each group consisted 40 patient then the severity of mastalgia in the three groups before, through and after intervention. Radiological assessment was done before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* all females with mastalgia aged 18 to 55

Exclusion Criteria:

Pregnant and lactating women, patient who had a recent breast abscess or breast drainage, patient used omega-3 and vitamin E supplementation before the trial and postmenopausal women.

-

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
improvement of pain severity | 3 months
  improvement of pain on visual analogue scale

SECONDARY OUTCOMES:
improvement of radiological finding | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Rehab Sabry, Cairo, Muslim, Egypt

IPD SHARING:
Plan to Share IPD: No